CLINICAL TRIAL: NCT06944977
Title: Early Childhood Caries Prevention: Effectiveness of Mother-Child Oral Health Care Programme (BASIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORKHAFIZAH SADDKI (Other)
Responsible Party: Sponsor-Investigator, NORKHAFIZAH SADDKI, ASSOCIATE PROFESSOR DR., Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00010568
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries
Keywords: anticipatory guidance; home visit; early childhood caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BASIS program (Experimental): Prenatal and postnatal anticipatory guidance with home visits
  Interventions: Behavioral: Anticipatory guidance and postnatal home visits
- Ministry of Health early childhood oral healthcare program (Active Comparator): Postnatal anticipatory guidance
  Interventions: Behavioral: Anticipatory guidance

INTERVENTIONS:
Behavioral: Anticipatory guidance and postnatal home visits — Anticipatory guidance to pregnant women, followed by scheduled home visits at 6, 12, and 18 months
  Arms: BASIS program
Behavioral: Anticipatory guidance — Postnatal anticipatory guidance
  Arms: Ministry of Health early childhood oral healthcare program

SUMMARY:
The goal of this two-arm, parallel-group cluster randomized controlled trial was to assess the effectiveness of the mother-child initiated oral health care program, termed BASIS, in preventing early childhood caries (ECC).

The main questions it aims to answer are:

* To compare mean knowledge and attitudes scores in the prevention of ECC among mothers of toddlers in the study group before and after receiving the BASIS program.
* To compare mean knowledge and attitude scores in the prevention of ECC between mothers of toddlers in the study group after receiving the BASIS program and mothers of toddlers in the control group after receiving the current Ministry of Health (MOH) programs.
* To compare oral health care practices in the prevention of ECC between mothers in the study group after receiving the BASIS program and mothers in the control group after receiving the current MOH program.
* To compare caries incidence between toddlers in the study group and toddlers in the control group after mothers' exposure to the BASIS program and the current MOH program, respectively.

Researchers will compare the BASIS program to the MOH program to see if the BASIS is effective to prevent ECC.

Participants of the BASIS program:

* Received anticipatory guidance delivered during pregnancy and after given birth at 6 months and 12 months
* Complete self-administered questionnaires measuring the knowledge, attitudes and practices related to the prevention of ECC during pregnancy and after given birth at 6 months, 12 months and 18 months
* Have their child oral cavity clinically examined at 6 months, 12 months and 18 months

ELIGIBILITY:
Inclusion Criteria:

* First-time pregnant women
* Aged 18 years and above
* In their third trimester
* Singleton pregnancy
* Able to read and write in Malay language
* Own a mobile phone with WhatsApp
* Will be the primary caretaker of their newborn

Exclusion Criteria:

• Diagnosed with cognitive disorders

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study enrolled pregnant women. Therefore, only females are eligible to participate
Enrollment: 154 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Changes in dental caries experience of the children from the age of 6 month to 18 months | From the age of 6 month to 18 months
  All surfaces of the four upper and lower front teeth of the children were examined at three time points: when the child reached 6 months old, 12 months old, and 18 months old. A sound tooth with no evidence of caries was coded as 0, while a tooth with evidence of caries, whether non-cavitated (such as white or brown spot lesions) or cavitated, was coded as 1.

SECONDARY OUTCOMES:
Change in knowledge, attitudes, and practices of mothers regarding the prevention of ECC assessed by self-administered questionnaire from enrollment to the end of the intervention at 18 months postpartum | From enrollment to the end of the intervention at 18 months postpartum
  The knowledge section of the questionnaire includes 30 items with responses in a close-ended format (true, false, and do not know). Correct answers receive 1 mark, while incorrect and 'do not know' responses receive no marks, resulting in a total score ranging from 0 to 30, with higher scores indicating better knowledge. The attitude domain consists of 12 items rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), with negatively worded statements re-coded in reverse. The total attitude scores range from 12 to 60, with higher scores reflecting a more positive attitude. The practices domain includes 21 items, with most questions using a yes or no response. Two items-feeding the child sweet food and cleaning the child's mouth/teeth in a day in a week-are assessed on a frequency scale. Responses for each practice item are described in terms of frequency and percentage, rather than being numerically scored and summed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tudan Health Clinic, Miri, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No
Ethical considerations